CLINICAL TRIAL: NCT05625997
Title: Intravascular Lithotripsy Plus Drug-coated Balloon in Calcified Small Coronary Vessels: a Feasibility Exploratory Study
Brief Title: Shockwave IVL + DCB
Status: Recruiting | Type: Observational
Sponsor: Rede Optimus Hospitalar SA (Network)
Responsible Party: Sponsor
Other Study IDs: RO-220203
Record Dates: First submitted 2022-11-15; First posted 2022-11-23 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Calcified Lesions in Small Coronary Vessels

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Drug-eluting stent (DES) implantation as interventional strategy for lesions in small coronary arteries is the current standard of care in many centers worldwide, but is associated with increased risk of late treatment failure in small vessels, as compared with larger coronary arteries. Randomized and observational studies have been shown that coronary intervention with drug-coated balloons (DCB) provide a promising alternative to DES implantation in small vessels, while avoiding the risk of a permanent vascular implant. Furthermore, lesions in small vessels are frequently concomitant with diffuse disease and/or distal location, where the presence of calcification is an additional common feature. Intravascular lithotripsy (IVL) has been recently introduced as a novel adjunctive technology to treat calcified lesions.

This study will explore the hypothesis that IVL has the potential to enhance the results of coronary balloon dilatation of small vessels with calcified lesions, therefore increasing the likelihood of optimal DBC intervention.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or older
2. Coronary artery disease with percutaneous intervention clinically indicated to treat one or more lesions fulfilling all criteria below:

   * De novo lesion with diameter stenosis > 50% (visual analysis)
   * Coronary vessel diameter < 3.0 mm (visual analysis)
   * Severe calcification at the target segment, defined as fluoroscopic radiopacities noted without cardiac motion prior to contrast injection involving both sides of the arterial wall in at least 1 location OR Intravascular Ultrasound/Optical Coherence Tomography (IVUS/OCT) demonstrated calcium angle of ≥270° on at least 1 cross section.
3. Written informed consent

Exclusion Criteria:

1. Previous coronary intervention at or < 10 mm distant from target segment at any time.
2. Lesion length ≥ 40 mm.
3. Planned atherectomy or cutting/scoring balloon use.
4. Bifurcation lesion.
5. Thrombus containing lesion.
6. Life expectancy < 12 months due to other co-morbid condition(s) that could limit patient's ability to participate in clinical study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a diminished blood flow in their calcified small coronary vessels
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-06-16 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Successful IVL plus DCB | at 1 month follow-up
  Successful IVL plus DCB in the absence of target lesion failure (TLF);
  "Successful IVL plus DCB" will be defined as a composite of:
  * IVL application at the target site, AND
  * DCB inflation at the target site, AND
  * Residual in-segment diameter stenosis <40% by quantitative coronary angiography, in the absence of final serious angiographic complications (≥ Grade D dissection, perforation, abrupt closure, final TIMI flow ≤ II), AND
  * Without the need for bailout scoring/cutting balloon or atherectomy-based strategy, AND
  * Without the need for bailout stenting.
  TLF will be defined as a composite of clinically driven revascularization, OR myocardial infarction, OR cardiac death related to the target lesion.

CONTACTS AND LOCATIONS:
Overall Officials: Flavio Ribichini, MD, Principal Investigator — Universita di Verona; Pedro Lemos, MD, Principal Investigator — Hospital Israelita Albert Einstein, São Paulo
Locations (2):
- Hospital Israelita Albert Einstein, São Paulo, Brazil
- University of Verona, Verona, Italy